CLINICAL TRIAL: NCT03511690
Title: Testing an Intelligent Tutoring System Intervention to Enhance Genetic Risk Assessment in Underserved Blacks and Latinas at Risk of Hereditary Breast Cancer
Brief Title: Testing an Intelligent Tutoring System to Enhance Genetic Risk Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Virginia Commonwealth University (Other); Cornell University (Other)
Responsible Party: Principal Investigator, Alejandra Hurtado de Mendoza, Assistant Professor, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1R21NR016905-01A1 (NIH)
Record Dates: First submitted 2018-04-16; First posted 2018-04-30 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Hereditary Breast and Ovarian Cancer
Keywords: Latinas, African Americans
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Intervention Model Description: Participants are randomized to an immediate or delayed arm
Who Masked: Outcomes Assessor
Masking Description: Randomization schedules will be developed by the biostatistician and administered by an individual (staff) not involved in the study analyses so that the statistician will be blinded to the allocation. This method will ensure unbiased results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate BRCA-Gist Intervention (Experimental): Participants randomized to immediate BRCA-gist will complete the adapted intervention and immediately complete a baseline survey. They will be asked to complete a second survey two weeks after completion of the first one. BRCA-gist is a web-based tutoring system that emulates one-to-one human tutoring via avatars to communicate risk of BRCA1/2. We estimate a completion time of 90 minutes.
  Interventions: Behavioral: BRCA-Gist
- Delayed BRCA-Gist Intervention (Experimental): Participants randomized to delayed BRCA-gist will initially complete a baseline survey. Two weeks after completion of that survey, they will complete the adapted intervention and immediately complete a second survey.
  Interventions: Behavioral: BRCA-Gist

INTERVENTIONS:
Behavioral: BRCA-Gist — BRCA-gist is an innovative Intelligent Tutoring System intervention that uses avatars to emulate tailored one-to-one human tutoring and includes the bottom-line meaning of risk messages. BRCA-gist is designed to provide the same information contained in four modules from the NCI webpages: "breast cancer and metastasis," "risk factors," "genetic mutation testing," and "the consequences of testing.

SUMMARY:
Participating in genetic cancer risk assessments (GCRA) for hereditary breast and ovarian cancer can inform treatment and risk management decisions and improve breast cancer outcomes. However, Latina and Black women underuse GCRA services, which may increase breast cancer disparities. This study will adapt and test the impact of an easily scalable novel Tutoring System intervention to enhance GCRA use and improve psychosocial outcomes in a clinical sample of underserved Latina and Black women at risk of hereditary breast and ovarian cancer.

DETAILED DESCRIPTION:
Specific Aims BRCA1/2 mutations are the most commonly identified Hereditary Breast and Ovarian Cancer (HBOC) mutations. Women with these mutations have a 50-80% lifetime risk of developing breast cancer. Breast cancer survivors with a BRCA1/2 mutation are at a higher risk of developing contralateral breast cancer than survivors without mutations. The National Comprehensive Cancer Network (NCCN) recommends referral for HBOC genetic cancer risk assessments (genetic counseling and consideration of genetic testing for a single gene or panel testing; GCRA) for women at high risk for carrying a mutation. Obtaining a positive test can inform treatment in newly diagnosed breast cancer patients and management in survivors and unaffected women. Unfortunately, Latina and Black women have lower GCRA use than non-Latina Whites. Reasons for lower GCRA use include access and psychosocial factors (e.g. low knowledge, medical mistrust, low health literacy, anticipated negative emotions). There have been few GCRA interventions in ethnic minorities; two recent efforts largely focused on improving access, awareness, and knowledge with mixed success of impacting uptake. Theoretically guided interventions that support GCRA uptake in underserved populations are needed. Intervention development is particularly important given the growing complexity of multiplex gene testing and the potential to identify founder mutations or large rearrangements that are more prevalent in specific ethnic groups.

Our preliminary data with at-risk Black and Latina women suggests that improving access does not necessarily translate into higher GCRA uptake and that providers face challenges in communicating HBOC risk information. Patients have difficulty understanding HBOC numerical risk information, especially populations with low health literacy. Additionally, many existing educational tools were not theoretically derived, tend to prioritize quantitative risk communication, and do not often consider emotional aspects, despite evidence that emotions influence risk perceptions. Fuzzy Trace Theory posits that rather than relying on factual knowledge and quantitative risk comprehension, people construct gist representations that are anchored on culture and capture the essential bottom-line meaning of risk information, including the emotional experience. Informed by Fuzzy Trace Theory, BRCA-gist is an innovative Intelligent Tutoring System intervention that uses avatars to emulate tailored one-to-one human tutoring and includes the bottom-line meaning of risk messages. The preliminary efficacy of BRCA-gist was established in an experimental laboratory setting with mostly non-Hispanic White college students. Adapting BRCA-gist for a clinical sample of ethnically/racially diverse women at increased risk of carrying a mutation is important. Thus, BRCA-gist constitutes a scalable, inexpensive intervention with promising translational applications and potential to reduce disparities.

The goal of this mixed methods study is to adapt BRCA-gist and test the feasibility, acceptability, and efficacy of this innovative intervention in a sample of Black and Latina women at risk of HBOC (based on NCCN criteria using personal and family history of cancer). Using the Learner Verification and Revision framework, in Aim 1 we will gather input from site staff and community providers (n=10) about adaptations for implementation in clinical settings and from at-risk Latina and Black women (n=20) about cultural adaptations. In Aim 2 we will test the feasibility, acceptability, and efficacy of the adapted BRCA-gist on uptake of GCRA services. We will recruit 50 women nationally. After completing a brief baseline survey, we will randomize participants to an immediate intervention arm or a delayed arm. Women will complete a baseline survey and a two-week follow up survey. Primary outcomes include change in knowledge, attitudes, and intention about GCRA from baseline to follow-up

Aim 1: Adapt BRCA-gist. Providers and at-risk Black and Latina women will do the BRCA-gist intervention and provide feedback and suggestions to make cultural adaptations to implement BRCA-gist in community/clinic settings.

Aim 2: Test the feasibility, acceptability, and efficacy of BRCA-gist intervention in a delayed intervention trial.

H.2.1. We expect high overall retention (≥75%). H.2.2. We expect high satisfaction among women in the BRCA-gist arm (≥75%). H.2.3. Participants will have a greater increase in knowledge, gist comprehension, and intentions to use GCRA after attending to BRCA-Gist compared to the delayed arm.

H.2.4. Participants will have a higher uptake of GCRA services 2 weeks after they attend to BRCA-Gist compared to the delayed arm.

This project builds on our interdisciplinary teams' expertise in using innovative technologies to improve risk communication, disparities, translational genomics, cancer control interventions, and emotions. If successful, BRCA-gist can be tested in larger samples and could easily be disseminated into clinical settings and community clinics that serve underserved populations at increased risk for cancer.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black and/or Latina
* English proficiency
* Be 18 years old or older
* Be able to provide informed consent
* Be at risk of carrying HBOC mutation using personal/family cancer histories based on the NCCN guidelines

Exclusion Criteria:

* Prior participation in genetic counseling or genetic testing for hereditary cancer risk.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 95 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Breast Cancer Genetics Knowledge | Aim 2. From baseline to two week after the baseline.
  Breast cancer genetics knowledge will be assessed with 13-items from Erblich and colleagues' scale where participants evaluate whether statements about breast cancer genetics are true or false. The numbers of correct responses are added to create a score ranging from 0-13. Higher scores mean higher breast cancer genetics knowledge.
Intentions to participate in genetic counseling | Aim 2. From baseline to two week after the baseline.
  Intentions to participate in genetic councSussner, Jandorf, Thompson, and Valdimarsdottir, 2010)
Perceived pros and cons of genetic counseling and testing | Aim 2. From baseline to two week after the baseline.
  Perceived pros and cons of genetic counseling and testing will be measured with a13-item 5-response Likert-type scale from Thompson and colleagues (2000) where participants rate their degree of agreement with statements about the potential benefits (7 items) and concerns of undergoing GCT (5 items). The cons items are reverse coded. Items are summed. Higher score means higher perceived positive attitudes. Scores range from 13-65.

SECONDARY OUTCOMES:
Uptake of Genetic Counseling | Two weeks after the intervention
  Scale
Self-efficacy about participating in genetic counseling | within one hour before the intervention and within one hour post-intervention
  Self-efficacy about participating in genetic counseling will be measured with the Genetic Testing and Counseling Self-efficacy Scale (Hendy, Lyons, Breakwell, 2006). The scale includes 3 items on a 5-point Likert-type response scale ranging from "completely agree" to "completely disagree." Items are summed. Scores range from 3-15. Higher scores indicate higher self-efficacy in participating in counseling and testing.
Emotions about developing breast cancer and about participating in genetic counseling | within one hour before the intervention and within one hour post-intervention
  Emotion about participating in genetic counseling will be assessed with Andersen's (2003) 5 item scale that captures scale to assess individuals' worry about developing breast cancer and with Caballero's (2007) scale scale to measure anticipatory emotions (how participants feel right now about participating in GCRA services in the future). Participants will report whether they feel positive (e.g. relief) and negative anticipatory emotions (e.g. worry) (Yes/No) and the level of intensity on a 7-point Likert-scale
Health Literacy and Numeracy | within one hour before the intervention
  General health literacy and numeracy with the Test of Functional Health Literacy in Adults (S-TOFHLA) short version that includes four numeracy items and two prose passages (Baker et al., 1999).
Mistrust about the medical system | within one hour before the intervention
  Mistrust about the medical system will be measured with the 7-item Medical Mistrust Index (Laveist et al., 2009)
Declarative Knowledge of Breast Cancer, Genetic Testing, and Genetic Risk | within one hour before the intervention and within one hour post-intervention
  Declarative Knowledge of Breast Cancer, Genetic Testing, and Genetic Risk - This scale developed by Wolfe and colleagues (2014) includes 52 four-alternative multiple-choice items about knowledge about breast cancer, genetic risk, and genetic testing. The percentage of correct answers are calculated. Higher percentages mean higher knowledge
Gist Comprehension of Genetic Cancer Risk | within one hour before the intervention and within one hour post-intervention
  Gist Comprehension of Genetic Cancer Risk (30 items). We will measure Gist Comprehension of Genetic Cancer Risk with a scale developed by Wolfe et al (2014). This 30-item Likert-type scale assesses gist comprehension of key information on breast cancer and genetic testing. The scale ranges from 1-7 (ranging from strongly disagree to strongly agree with correct responses). Responses are averaged. Higher scores indicate higher gist comprehension.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra H Hurtado de Mendoza, PhD, Principal Investigator — Georgetown University; Vanessa Sheppard, PhD, Principal Investigator — Virginia Commonwealth University
Locations (4):
- United States (4):
  - Capital Breast Care Center, Washington D.C., District of Columbia
  - Georgetown University, Washington D.C., District of Columbia
  - Nueva Vida, Alexandria, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Background] Easton DF. How many more breast cancer predisposition genes are there? Breast Cancer Res. 1999;1(1):14-7. doi: 10.1186/bcr6. Epub 1999 Aug 23. No abstract available. PMID 11250676
- [Background] Chen S, Parmigiani G. Meta-analysis of BRCA1 and BRCA2 penetrance. J Clin Oncol. 2007 Apr 10;25(11):1329-33. doi: 10.1200/JCO.2006.09.1066. PMID 17416853
- [Background] Malone KE, Begg CB, Haile RW, Borg A, Concannon P, Tellhed L, Xue S, Teraoka S, Bernstein L, Capanu M, Reiner AS, Riedel ER, Thomas DC, Mellemkjaer L, Lynch CF, Boice JD Jr, Anton-Culver H, Bernstein JL. Population-based study of the risk of second primary contralateral breast cancer associated with carrying a mutation in BRCA1 or BRCA2. J Clin Oncol. 2010 May 10;28(14):2404-10. doi: 10.1200/JCO.2009.24.2495. Epub 2010 Apr 5. PMID 20368571
- [Background] Kauff ND, Satagopan JM, Robson ME, Scheuer L, Hensley M, Hudis CA, Ellis NA, Boyd J, Borgen PI, Barakat RR, Norton L, Castiel M, Nafa K, Offit K. Risk-reducing salpingo-oophorectomy in women with a BRCA1 or BRCA2 mutation. N Engl J Med. 2002 May 23;346(21):1609-15. doi: 10.1056/NEJMoa020119. Epub 2002 May 20. PMID 12023992
- [Background] Levy DE, Byfield SD, Comstock CB, Garber JE, Syngal S, Crown WH, Shields AE. Underutilization of BRCA1/2 testing to guide breast cancer treatment: black and Hispanic women particularly at risk. Genet Med. 2011 Apr;13(4):349-55. doi: 10.1097/GIM.0b013e3182091ba4. PMID 21358336
- [Background] Glenn BA, Chawla N, Bastani R. Barriers to genetic testing for breast cancer risk among ethnic minority women: an exploratory study. Ethn Dis. 2012 Summer;22(3):267-73. PMID 22870568
- [Background] Sussner KM, Jandorf L, Thompson HS, Valdimarsdottir HB. Barriers and facilitators to BRCA genetic counseling among at-risk Latinas in New York City. Psychooncology. 2013 Jul;22(7):1594-604. doi: 10.1002/pon.3187. Epub 2012 Sep 16. PMID 22987526
- [Background] Sussner KM, Edwards T, Villagra C, Rodriguez MC, Thompson HS, Jandorf L, Valdimarsdottir HB. BRCA genetic counseling among at-risk Latinas in New York City: new beliefs shape new generation. J Genet Couns. 2015 Feb;24(1):134-48. doi: 10.1007/s10897-014-9746-z. Epub 2014 Aug 15. PMID 25120034
- [Background] Thompson HS, Valdimarsdottir HB, Jandorf L, Redd W. Perceived disadvantages and concerns about abuses of genetic testing for cancer risk: differences across African American, Latina and Caucasian women. Patient Educ Couns. 2003 Nov;51(3):217-27. doi: 10.1016/s0738-3991(02)00219-7. PMID 14630378
- [Background] Armstrong K, Micco E, Carney A, Stopfer J, Putt M. Racial differences in the use of BRCA1/2 testing among women with a family history of breast or ovarian cancer. JAMA. 2005 Apr 13;293(14):1729-36. doi: 10.1001/jama.293.14.1729. PMID 15827311
- [Background] Mays D, Sharff ME, DeMarco TA, Williams B, Beck B, Sheppard VB, Peshkin BN, Eng-Wong J, Tercyak KP. Outcomes of a systems-level intervention offering breast cancer risk assessments to low-income underserved women. Fam Cancer. 2012 Sep;11(3):493-502. doi: 10.1007/s10689-012-9541-7. PMID 22711611
- [Background] Ricker C, Lagos V, Feldman N, Hiyama S, Fuentes S, Kumar V, Gonzalez K, Palomares M, Blazer K, Lowstuter K, MacDonald D, Weitzel J. If we build it ... will they come?--establishing a cancer genetics services clinic for an underserved predominantly Latina cohort. J Genet Couns. 2006 Dec;15(6):505-14. doi: 10.1007/s10897-006-9052-5. PMID 17106633
- [Background] Hall MJ, Olopade OI. Disparities in genetic testing: thinking outside the BRCA box. J Clin Oncol. 2006 May 10;24(14):2197-203. doi: 10.1200/JCO.2006.05.5889. PMID 16682739
- [Background] Weitzel JN, Clague J, Martir-Negron A, Ogaz R, Herzog J, Ricker C, Jungbluth C, Cina C, Duncan P, Unzeitig G, Saldivar JS, Beattie M, Feldman N, Sand S, Port D, Barragan DI, John EM, Neuhausen SL, Larson GP. Prevalence and type of BRCA mutations in Hispanics undergoing genetic cancer risk assessment in the southwestern United States: a report from the Clinical Cancer Genetics Community Research Network. J Clin Oncol. 2013 Jan 10;31(2):210-6. doi: 10.1200/JCO.2011.41.0027. Epub 2012 Dec 10. PMID 23233716
- [Background] Graves KD, Christopher J, Harrison TM, Peshkin BN, Isaacs C, Sheppard VB. Providers' perceptions and practices regarding BRCA1/2 genetic counseling and testing in African American women. J Genet Couns. 2011 Dec;20(6):674-89. doi: 10.1007/s10897-011-9396-3. Epub 2011 Aug 6. PMID 21822773
- [Background] Wolfe CR, Reyna VF, Widmer CL, Cedillos EM, Fisher CR, Brust-Renck PG, Weil AM. Efficacy of a web-based intelligent tutoring system for communicating genetic risk of breast cancer: a fuzzy-trace theory approach. Med Decis Making. 2015 Jan;35(1):46-59. doi: 10.1177/0272989X14535983. Epub 2014 May 14. PMID 24829276
- [Background] Zikmund-Fisher BJ, Fagerlin A, Ubel PA. Risky feelings: why a 6% risk of cancer does not always feel like 6%. Patient Educ Couns. 2010 Dec;81 Suppl:S87-93. doi: 10.1016/j.pec.2010.07.041. Epub 2010 Aug 23. PMID 20739135
- [Background] Reyna VF, Nelson WL, Han PK, Pignone MP. Decision making and cancer. Am Psychol. 2015 Feb-Mar;70(2):105-18. doi: 10.1037/a0036834. PMID 25730718
- [Background] Caballero A, Carrera P, Munoz D, Flor S. Emotional ambivalence in risk behaviors: the case of occasional excessive use of alcohol. Span J Psychol. 2007 May;10(1):151-8. doi: 10.1017/s1138741600006417. PMID 17549888
- [Background] Baker DW, Williams MV, Parker RM, Gazmararian JA, Nurss J. Development of a brief test to measure functional health literacy. Patient Educ Couns. 1999 Sep;38(1):33-42. doi: 10.1016/s0738-3991(98)00116-5. PMID 14528569
- [Background] Sheppard VB, Mays D, LaVeist T, Tercyak KP. Medical mistrust influences black women's level of engagement in BRCA 1/2 genetic counseling and testing. J Natl Med Assoc. 2013 Spring;105(1):17-22. doi: 10.1016/s0027-9684(15)30081-x. PMID 23862292
- [Background] LaVeist TA, Isaac LA, Williams KP. Mistrust of health care organizations is associated with underutilization of health services. Health Serv Res. 2009 Dec;44(6):2093-105. doi: 10.1111/j.1475-6773.2009.01017.x. Epub 2009 Sep 2. PMID 19732170
- [Background] Erblich J, Brown K, Kim Y, Valdimarsdottir HB, Livingston BE, Bovbjerg DH. Development and validation of a Breast Cancer Genetic Counseling Knowledge Questionnaire. Patient Educ Couns. 2005 Feb;56(2):182-91. doi: 10.1016/j.pec.2004.02.007. PMID 15653247
- [Background] Hendy J, Lyons E, Breakwell GM. Genetic testing and the relationship between specific and general self-efficacy. Br J Health Psychol. 2006 May;11(Pt 2):221-33. doi: 10.1348/135910705X52543. PMID 16643695